CLINICAL TRIAL: NCT02402413
Title: Ultrasound Three-dimensional Characterization of Ovarian Morphology in Women With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate professor, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCOSCA
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: PCOS; Hyperandrogenism
MeSH Terms: conditions — Hyperandrogenism | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCOS women (Experimental)
  Interventions: Procedure: Ultrasound; Procedure: Determination of concentrations of androgens; Device: Three dimensional ultrasound probe

INTERVENTIONS:
Procedure: Ultrasound — The patients will be subjected to ultrasound bi-dimensional or three-dimensional. Will Be calculated the ratio stroma/volume with both methods
  Other Names: Ultrasound evaluation of ovarian morphology
Procedure: Determination of concentrations of androgens — Determination of concentrations of serum levels of circulating androgens
Device: Three dimensional ultrasound probe — Capture of ovarian three dimensional volumes

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common endocrine disorders occurring in women of reproductive age. PCOS is considered a syndrome of ovarian dysfunction that is characterized by the heterogeneous clinical manifestation of infrequent or absent menstrual cycles, hyperandrogenism, and polycystic ovarian morphology.

An important ultrasound parameter is the ratio stroma/ovary, the ratio of the volume, evaluated in two-dimensional ultrasound, of the stroma, that secrete androgen, and the ovary. It has been shown that when this ratio is higher than a third the levels of circulating androgens and high. Aim of the present study is to assess whether this ratio, determined with three-dimensional ultrasound, is correlated to the increase of androgens.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of infrequent or absent menstrual cycles and/or PCOS ultrasound feature and/or clinical or biochemical hyperandrogenism
* Did not take hormonal contraception, fertility therapies, or insulin sensitizers in the three months prior to enrollment

Exclusion Criteria:

* Pregnancy

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Androgens serum levels in women with ultrasound morphological PCO | up to 1 year

REFERENCES:
- [Result] Fulghesu AM, Ciampelli M, Belosi C, Apa R, Pavone V, Lanzone A. A new ultrasound criterion for the diagnosis of polycystic ovary syndrome: the ovarian stroma/total area ratio. Fertil Steril. 2001 Aug;76(2):326-31. doi: 10.1016/s0015-0282(01)01919-7. PMID 11476780